CLINICAL TRIAL: NCT03333434
Title: Effectiveness of Ankle-7 Orthosis vs HAFO Orthosis on Gait Performance in Diplegic Cerebral Palsied Children
Brief Title: Effectiveness Ankle-7 Orthosis VS HAFO Orthosis on Gait in Diplegic CPChildren
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: Otto Bock Healthcare Products GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UDGEE_2012_OTTObock
Record Dates: First submitted 2017-10-02; First posted 2017-11-07 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2017-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- AFO - Ankle_7 group (Other): AFO is active comparator, ANKLE7 is the experimental treatment
  Interventions: Device: Carbon Ankle Seven spring (A7 - Otto Bock, Germany); Device: Hinged AFO
- Ankle-7 - AFO group (Other): AFO is active comparator, ANKLE7 is the experimental treatment
  Interventions: Device: Carbon Ankle Seven spring (A7 - Otto Bock, Germany); Device: Hinged AFO

INTERVENTIONS:
Device: Carbon Ankle Seven spring (A7 - Otto Bock, Germany)
Device: Hinged AFO

SUMMARY:
Ankle foot orthoses (AFO) are frequently used to improve locomotor skills of cerebral palsied children (CP) although the level of scientific evidence to support their use is still moderate. Carbon Ankle Seven spring (A7 - Otto Bock, Germany) is specifically designed to store energy when loaded and release it at toe-off in order to improve gait performance with respect to non-energy-storing AFOs. The aim of this work is to verify the superiority of the ankle-7 orthosis compared to the more widespread AFO, to improve the functionality and walking function of children with spastic diplegia and PCI.

DETAILED DESCRIPTION:
The project is divided into the following phases:

T0 - at the beginning of the study children included will be subject to the following procedures and assessments:

1. demographic and anthropometric data collection;
2. randomization by concealed allocation to one of the following two groups:

   * AFO - Ankle_7 group
   * Ankle-7 - AFO group Both, AFO and ankle-7, will be tailored to the patient

   The two groups are distinguished by the order of the assignment of the two orthoses, respectively defined as the first assignment orthosis (O_1) and second assignment orthosis (O_2). The first group will use the orthoses AFO as a first assignment and then the orthoses Ankle_7, while the second group will use the two orthoses according to the reverse order. The two will be used with the same orthotic footwear, with the exception of the cases where it will be necessary to change it due to accretion.
3. collection of the measures necessary for making the two orthotic devices at OttoBock of Reggio Emilia
4. training in the use of the orthoses according to a standardized protocol;
5. try on the patient's in-process first assignment orthoses (O_1) and subsequent delivery of them (see Annex A);

Subsequently, the patient will use O_1 for a period of 4-6 weeks.

T1 - patients will receive the following procedures and assessments:

1. try on the patient's in-process second assignment orthoses (O_2)
2. instrumental gait analysis and video recording of the walking while using O_1 (covered by elastic gaiters);
3. withdrawal of O_1
4. delivery of O_2 to the patient

Subsequently, the patient will use O_2 for a period of 4-6 weeks.

T2 - patients will undergo the following procedures and evaluations:

1. instrumental gait analysis and video recording of the walking while using O_2 (covered by elastic gaiters);
2. return of O_1 to the patient;
3. Delivery of the diaries and directions for completing and mailing back them at the end of the follow-up period;

T3 - three months follow-up to detect the preference of use of AFO or Ankle-7 (by the child/parent)

ELIGIBILITY:
Inclusion Criteria:

* - Clinical indication to the use of orthoses to improve the walking function confirmed by instrumental parameters obtained from analysis of the path (dynamic electromyography, optoelectronic stereophotogrammetry analysis);
* Patients who already have AFO orthoses (or ankle-7) that need to be renewed;
* Patients with new clinical indication to the use of orthoses but not yet in possession of the same;
* Informed consent from parents / guardians of the child

Exclusion Criteria:

* Cognitive disabilities that may affect the child's participation in the activities related to this study, in the opinion of the investigators;
* Lower limbs sensory disability that may affect any beneficial effects of the use of the orthoses, in the opinion of the investigators;
* Other diseases associated or not associated with PCI that, according to investigators, could affect the child's participation in the activities related to this study (eg: drug-resistant epilepsy);
* Administration of antispasmodic drugs in the last 6 months;
* Functional surgery of the lower limbs in the last 6 months;
* Indication for surgical treatment to be carried out within 6 months after the date of inclusion in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11-30 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Change from right and left ankle joints power generation in stance phase after the use of first orthosis to right and left ankle joints power generation in stance phase after the use of second orthosis | After a 4-6 week period of use of first orthosis and after a 4-6 week period of use of second orthosis
  Measured by instrumental gait analysis (ratio of watt to kilogram)

SECONDARY OUTCOMES:
knee joint kinematics | After a 4-6 week period of use of first orthosis and after a 4-6 week period of use of second orthosis
  average extension in degrees of the right and left knees during initial contact, loading response and mid-stance measured by instrumental gait analysis
stride length | After a 4-6 week period of use of first orthosis and after a 4-6 week period of use of second orthosis
  stride length right and left leg, measured by instrumental gait analysis (percentage of height)
walking speed | After a 4-6 week period of use of first orthosis and after a 4-6 week period of use of second orthosis
  walking speed measured by instrumental gait analysis (ratio of percentage of height to seconds)
preference of use of AFO or Ankle_7 | After a 4-6 week period of use of first orthosis, after a 4-6 week period of use of second orthosis and after 3 months after three months when the child could freely use both orthoses
  determined from a self- compiled diary
clinical evaluation of the walking function | After a 4-6 week period of use of first orthosis and after a 4-6 week period of use of second orthosis
  Using video-recording of children during walking and the Visual Gait Assessment Scale (OGS). (Boyd R, Graham HK. 1999)

CONTACTS AND LOCATIONS:
Overall Officials: Adriano Ferrari, Principal Investigator — University of Modena and Reggio Emilia

DOCUMENTS (1):
  • Study Protocol (2013-09-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT03333434/Prot_000.pdf